CLINICAL TRIAL: NCT03362359
Title: An Open-label, Single-arm, Rater-blinded, Multicenter Phase 1/2 Study to Assess Safety and Diagnostic Accuracy and Radiotherapeutic Implications of Pre-operative Ga-68-PSMA-11 PET/CT Imaging in Comparison to Histopathology, in Newly-diagnosed Prostate Cancer (PCA) Patients at High Risk for Metastasis, Scheduled for Radical Prostatectomy (RP) With Extended Pelvic Lymph Node Dissection (EPLND)
Brief Title: Ga-68-PSMA-11 in High-risk Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: ABX CRO (Other); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ga-68-PSMA-11
Record Dates: First submitted 2017-10-18; First posted 2017-12-05 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: High-risk Prostate Cancer; Prostate Cancer; Prostate Cancer Metastatic; Lymphnode Metastasis
Keywords: prostatectomy; 68Ga-PSMA-11; EPLND
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ga-68-PSMA-11 (Experimental)
  Interventions: Drug: Ga-68-PSMA-11

INTERVENTIONS:
Drug: Ga-68-PSMA-11 — Single administration of 150 MBq (± 50 MBq), corresponding to a mass dose of ≤ 6 µg. A 2nd administration of 150 MBq (± 50 MBq), corresponding to a mass dose of ≤ 6 µg is possible in the unlikely case of a negative histological result (i.e. no prostate-specific membrane antigen (PSMA) expression in dissected lymph nodes) to verify if PSMA PET-positive tissue as seen on day 1 has not been removed during RP with EPLND.
  Other Names: 68Ga-DKFZ-PSMA; 68Ga-PSMA; 68Ga-PSMA(HBED); Glu-NH-CO-NH-Lys-(Ahx)-[68Ga(HBED-CC)]

SUMMARY:
This will be an open-label, single-arm, rater-blinded, multicenter, diagnostic phase 1/2 study to assess safety and diagnostic performance of Ga-68-PSMA-11 positron emission tomography / computer tomography (PET/CT) imaging to detect tumour tissue in patients with newly diagnosed PCA and a high risk for metastasis. As standard of truth, comprehensive histopathology covering prostate and the tributary pelvic lymph node system, will be used. Therefore, only patients scheduled for RP with EPLND (as part of their standard of care) will be eligible.

Patients will be recruited at up to 11 uro-oncological sites in Germany, Austria, and Switzerland, with access to a radiopharmaceutical laboratory, experienced to prepare 68Ga-labelled compounds, and high-quality PET/CT imaging. Upon histological confirmation of PCA, pre-operative staging will be performed according to European Association of Urology (EAU) guideline [Mottet et al. 2015] (to include pelvic MRI or CT and a 99mTc-bone scan), to establish the indication for RP with EPLND. If the indication is confirmed, patients will be invited to participate in the present study. After consenting, review of inclusion and exclusion criteria, as well as screening investigations will be performed by the uro-oncologist (day 0). Thereafter, patients are referred to the collaborating nuclear medicine department for tracer injection, imaging, and post-dose safety evaluations (day 1). Subsequent investigations (day 2 and at end of study) will be made by the uro-oncologist or experienced nuclear medicine physician. Study participation ends on day 7. Routine surgery (RP with EPLND) will be performed after end of study, but no later than 42 days after study inclusion. This sequence allows adequate characterisation of tracer safety, while at the same avoiding unnecessary delay of, or confounding safety signals from therapy.

In total, 150 evaluable patients will be included to receive a single 68Ga dose of 150 MBq (± 50 MBq), administered as i.v. infusion. Due to an assumed dropout rate of 15%, up to 173 patients will be included in study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male ≥ 18 years of age.
3. Histologically confirmed adenocarcinoma of the prostate.
4. High risk for metastasis, defined by either:

   1. stadium cT3 according to TNM (primary tumor, regional nodes, metastasis) Classification of Malignant Tumours (TNM), or
   2. Gleason Score >7, or
   3. Prostate-Specific Antigen (PSA) >20 ng/mL.
5. Patient scheduled for radical prostatectomy (RP) with extended pelvic lymph node dissection (EPLND) according to current guidelines 7 - 60 days after start of study.
6. Consent to practise contraception until end of study (6 days after Ga-68-PSMA-11 injection).
7. Preoperative PCA staging performed according to guidelines, to include a mandatory 99mTc bone scintigraphy and an optional pelvic MRI or CT, not older than 56 days prior to inclusion, according to standard of care.

Exclusion Criteria:

1. Known hypersensitivity to Ga-68-PSMA-11 or its components.
2. Presence of known lymph node metastases outside surgical field.
3. More than 5 bone metastases, as determined by 99mTc bone scintigraphy.
4. Previous prostate cancer therapy.
5. Administration of any kind of PET tracer within a period corresponding to 8 half-lives of the respective radionuclide.
6. Any other investigational medicinal product within 30 days prior and 7 days after receiving study medication.
7. Evidence of neuroendocrine small cell carcinoma.
8. Subjects not able to declare meaningful informed consent on their own (e.g. with legal guardian for mental disorders).
9. Simultaneous participation in other clinical trials

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male with prostate cancer
Enrollment: 173 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
True positive fraction (TPF) and false positive fraction (FPF) of identified tumour tissue in soft tissue, analysed separately for prostate gland and pelvic lymph nodes, using histopathology as standard of truth. | up to day 21
Frequency of occurrence and severity of abnormal findings in safety investigations (physical examination, vital signs, 12-lead ECG, pulse oximetry, clinical laboratory, adverse events, concomitant medication). | Day 0 - Day 7

SECONDARY OUTCOMES:
Number of identified bone lesions, per patient. | Day 1
Correlation coefficient of recovery-corrected standardized uptake values (SUV) plotted against Gleason score in primaries after RP | Day 1
Percentage of subjects for whom the RP and EPLND will not be conducted | Day 1
Quantity of circulating tumour cells in blood | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Giesel, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (8):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Germany (7):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Friedrich-Alexander-Universität Erlangen, Erlangen
  - Universität Duisburg-Essen, Essen
  - Albert-Ludwigs-Universität Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - Technische Universität München Klinikum rechts der Isar, München
  - Eberhard-Karls-Universität Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No